CLINICAL TRIAL: NCT02365714
Title: A Pilot Study of Stereotactic Accelerated Partial Breast Irradiation (SAPBI) for Post-Menopausal Women (>50 y/o) With Ductal Carcinoma in Situ (DCIS) or Early Stage Breast Cancer
Brief Title: CyberKnife Stereotactic Accelerated Partial Breast Irradiation (SAPBI)
Acronym: CK-SAPBI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC012015-02
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2016-06

CONDITIONS: Breast Cancer; DCIS; Invasive Ductal Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment-Radiation (Other): CyberKnife (CK) Stereotactic Accelerated Partial Breast Irradiation. Adjuvant radiation therapy delivered to the region around the lumpectomy cavity. Patients will receive 30 Gy in 5 fractions over 5-14 days.
  Interventions: Radiation: CK Stereotactic Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: CK Stereotactic Accelerated Partial Breast Irradiation — Adjuvant radiation therapy will be delivered to the region of the lumpectomy cavity once daily for 5 treatments over 5-10 days.
  Other Names: CyberKnife, SAPBI

SUMMARY:
This study will prospectively evaluate the technical feasibility, acute toxicity, late effects and oncologic outcomes of CyberKnife Stereotactic Accelerated Partial Breast Irradiation (CK-SAPBI) in early stage breast cancer. It will evaluate quality of life (QOL) issues as they relate to treatment-related side effects and cosmetic results.

DETAILED DESCRIPTION:
This study will determine the feasibility, acute and late toxicity as well as oncologic outcomes following CK-SAPBI.

ELIGIBILITY:
Inclusion Criteria:

* -Newly diagnosed Stage 0 or I breast cancer.
* On histological examination, the tumor must be DCIS or invasive non-lobular carcinoma of the breast
* Surgical treatment of the breast must have been wide excision, lumpectomy or partial mastectomy
* Age 50 years or greater
* ER positive: (≥1% of breast tumor cells express ER in their nuclei)
* PR (progesterone receptor) positive: (≥ 1% of breast tumor cells express PR in their nuclei)
* Her2 negative (IHC 0-1+; for IHC 2+, FISH (fluorescence in situ hybridization) must be non-amplified)
* Subjects with invasive tumors should undergo axillary sentinel lymph node evaluation or axillary lymph node dissection.
* Negative inked surgical margins of excision or re-excision, clear of invasive tumor (no cells on ink) and DCIS by at least 1 mm
* Negative post-excision or post-reexcision mammography if cancer presented with malignancy-associated microcalcifications with no remaining suspicious calcifications in the breast before radiotherapy. Alternatively, a specimen radiograph can be obtained showing all the suspicious calcifications.
* No involved axillary lymph nodes, N0(i+) allowed
* Enrollment and the plan to initiate of CyberKnife therapy within 12 weeks of the last breast cancer surgery.
* Target lumpectomy cavity/whole breast reference volume must be <30% based on treatment planning CT
* Signed study-specific informed consent form

Exclusion Criteria:

* -Patients with invasive lobular carcinoma or nonepithelial breast malignancies such as sarcoma or lymphoma.
* Patients with tumors greater than 2 cm
* Patients with surgical margins which cannot be microscopically assessed or not cleared by at least 2mm at pathological evaluation.
* Patients with multicentric carcinoma or with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy. Breast MRI will be recommended to exclude multicentric disease and additional suspicious areas will require biopsy to exclude malignancy.
* Patient with lymphovascular space invasion (LVSI).
* Patients with involved axillary nodes.
* Patients with collagen vascular diseases.
* Patient with known deleterious BRCA1/2 mutations or known mutations in other high penetrance genes (TP53, STK11, PTEN-phosphatase and tensin homolog, CDH1)
* Patients with prior ipsilateral breast irradiation.
* Patients with prior ipsilateral thoracic irradiation.
* Patients with Paget's disease of the nipple.
* Patients with diffuse suspicious microcalcifications.
* Patients with suspicious microcalcifications remaining on the post-excision mammogram.
* Patients receiving (neo)adjuvant systemic therapy other than hormonal therapy
* Patients with oncoplastic reconstruction and absence of surgical clips

Ages: 50 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Rudra, M.D., Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CyberKnife Arm: This is a single arm study for patients who are eligible for partial breast irradiation.
Period: Overall Study
Arm/Group | CyberKnife Arm
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 2 patients were enrolled. Age=55 and 63 at treatment. Race=African American in both.
Groups:
- CyberKnife Arm: Two patients were enrolled for CyberKnife. In one patient, the fiducials were unable to be tracked, so she received external beam partial breast irradiation.
Arm/Group | CyberKnife Arm
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 59 [55 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint for This Study is the Percentage of Enrolled Subjects in Whom CyberKnife SAPBI PBI is Technically Feasible to Deliver and Complete Treatment
Description: Only one of two patients were able to undergo CyberKnife SAPBI. We are measuring the percentage of enrolled subjects in whom CyberKnife SAPBI PBI is technically feasible to deliver and complete treatment
Time Frame: Enrollment to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Arm
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Feasibility
Description: How many patients were able to undergo CK SAPBI
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Arm
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Ipsilateral Breast Recurrence
Description: No patients have recurred to date.
Time Frame: 1 month post radiation treatment through 5 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Arm
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment-Radiation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-Radiation (N=2)
RT dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No